CLINICAL TRIAL: NCT03195374
Title: Assessment of the Prevalence of Analgesics Opioid Misuse in Chronic Non-cancer Pain Patients
Brief Title: Prescription Opioid Misuse Assessment
Acronym: POMA4
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CEIP-A Lyon (Unknown); CEIP-A Marseille (Unknown); CEIP-A Caen (Unknown); CEIP-A Lille (Unknown); CEIP-A Montpellier (Unknown); CEIP-A Nantes (Unknown); CEIP-A Poitiers (Unknown); CEIP-A Toulouse (Unknown); CEIP-A Bordeaux (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-338; 2016-A00648-43 (Other: 2016-A00648-43)
Record Dates: First submitted 2017-06-12; First posted 2017-06-22 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain
Keywords: Analgesic opioids; Misuse; Use disorder; Pain
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic non-cancer pain: Each addictovigilance centre will contact Pain Clinics in order to enroll patients meeting the inclusion criteria.
  Interventions: Other: Prescription Opioid Misus Index

INTERVENTIONS:
Other: Prescription Opioid Misus Index — Opioid misuse will be assessed by the Prescription Opioid Misuse Index (POMI) scale. A score ≥ 2 is considered positive and will define a misuse behavior.

SUMMARY:
Chronic pain is a worldwide health problem due to its high prevalence and its difficult management with a significant impact on quality of life. Pain and addiction co-occur frequently. Indeed, the prevalence of addiction in patients with chronic non-cancer pain may affect from 0% to 50% of patients (Højsted et al 2010). This large variability in the estimation of addiction prevalence in chronic non-cancer pain patients is at least partly due to a lack of standardization of the selected patients from the clinical or therapeutic point of view and the lack of consensus in the use of a specific evaluation tool or gold standard. Indeed, several tools are currently available at the international level with varying efficiencies and precisions (Chou et al 2009, Turk, Swanson, and Gatchel 2008, Højsted and Sjøgren 2007). In France, no data are available on the prevalence of analgesic opioid misuse in chronic non-cancer pain patients, due to the lack clinical studies and validated tools in French.

DETAILED DESCRIPTION:
This is an observational study . Each addictovigilance centre will contact Pain Clinics in order to enroll patients meeting the inclusion criteria. The questionnaires will be prepared and sent to the participating centres by the coordinating centre (Clermont-Ferrand). Participation in the study will be systematically proposed by the physician during the study inclusion period (3 months). Patients meeting all inclusion criteria will be enrolled after receiving oral information about the study.

This questionnaire can be semi-directed (doctor / nurse / CRA) and will be carried out during a consultation as part of their usual care. Answering the questionnaire should take no more than 10 minutes. No additional diagnostic or monitoring procedures will be applied to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) ≥ 18 years old
* Patients with chronic non-cancer pain for at least 6 months
* Patients treated with analgesic opioids for at least 3 months

Exclusion Criteria:

* Patients (male or female) < 18 years old
* Patients with chronic pain for less than 6 months
* Patients with cancer pain
* Patients treated with analgesic opioids for less than 3 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each addictovigilance centre will contact Pain Clinics in order to enroll patients meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 951 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Opioid misuse will be assessed by the Prescription Opioid Misuse Index (POMI) scale | at day 1
  A score ≥ 2 is considered positive and will define a misuse behavior

SECONDARY OUTCOMES:
Analgesic opioids used by the patient will be collected in the questionnaire | at day 1
Patients' profiles and associated risk factors of opioid misuse will be described through socio-demographic contained in the questionnaire | at day 1
  age, gender, family situation, employment status) and clinical data (type of pain, age of painful pathology, psychiatric comorbidities, abuse of other substances, etc

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas AUTHIER, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Derived] Kerckhove N, Delage N, Bertin C, Kuhn E, Cantagrel N, Vigneau C, Delorme J, Lambert C, Pereira B, Chenaf C, Authier N; Poma Network. Cross-sectional study of the prevalence of prescription opioids misuse in French patients with chronic non-cancer pain: An update with the French version of the POMI scale. Front Pharmacol. 2022 Sep 5;13:947006. doi: 10.3389/fphar.2022.947006. eCollection 2022. PMID 36133827